CLINICAL TRIAL: NCT00846079
Title: Myocardial Perfusion Assessment With Multidetector Computed Tomography
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tennessee Heart and Vascular Institute, P.C. (Other)
Collaborators: General Electric (Industry)
Responsible Party: Tracy Callister,MD, Tennessee Heart and Vascular Institute, P.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: THVI-101
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; stress testing
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Regadenoson (Lexiscan) [muti-detector computed tomography] — Regadenason, typical dosing
  Other Names: Lexiscan

SUMMARY:
Demonstrate the ability of muti-detector computed tomography to adequately perform stress testing will result in a veritable "one-stop shop" of non-invasive cardiac imaging that is, the ability to directly visualize heart arteries with high accuracy and to simultaniously determine the hemodynamic significance of any blockages visualized.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Adults undergoing myocardial perfusion SPECT imaging
* Adults with suspected coronary artery disease

Exclusion Criteria:

* Age <18
* Known or suspected renal insufficiency (Creatinine <1.7 mg/dl)
* Allergy to contrast
* Inability or contraindication to lexiscan or beta blocker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy (Sensitivity/Specificity/Positive Predictive Value/Negative Predictive Value) | 6 months

SECONDARY OUTCOMES:
Radiation dosimetry | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tennessee Heart and Vascular Institute, Hendersonville, Tennessee, United States